CLINICAL TRIAL: NCT04401384
Title: Effectiveness of Acupuncture and Doxylamine/Pyridoxine for Moderate to Severe Nausea and Vomiting in Pregnancy: A Randomized Controlled Two-by-two Factorial Trial
Brief Title: Effectiveness of Acupuncture and Doxylamine/Pyridoxine for Moderate to Severe Nausea and Vomiting in Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xiaoke Wu (Other)
Collaborators: Ningxia Hui Autonomous Region Hospital of TCM (Unknown); Jiangxi Maternal and Child Health Hospital (Other); Jixi Maternal and Child Health Hospital (Unknown); Luoyang Hospital of TCM (Unknown); Xuzhou Central Hospital (Other); First Affiliated Hospital of Heilongjiang Chinese Medicine University (Other); Shuangyashan Maternal and Child Health Hospital (Unknown); Heilongjiang provincial hospital (Unknown); Jiamusi Maternal and Child Health Hospital (Unknown); Hegang Maternal and Child Health Hospital (Unknown); Suihua Maternal and Child Health Hospital (Unknown); Mudanjaing Maternal and Child Health Hospital (Unknown); Affiliated Hospital of Jiamusi Medical University (Unknown)
Responsible Party: Sponsor-Investigator, Xiaoke Wu, Director of obstetrics and Gynecology Department, Heilongjiang University of Chinese Medicine
Organization: Heilongjiang University of Chinese Medicine (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NVPAct
Record Dates: First submitted 2020-05-18; First posted 2020-05-26 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Nausea and Vomiting of Pregnancy
Keywords: Nausea and Vomiting of Pregnancy; PUQE; Acupuncture; Diclectin
MeSH Terms: conditions — Nausea | interventions — dicyclomine, doxylamine, pyridoxine drug combination

STUDY DESIGN:
Intervention Model Description: Two by two factorial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Diclectin plus active acupuncture (Other): Diclectin (combination of doxylamine succinate (10 mg) and pyridoxine hydrochloride (10 mg) , 2-4 tablets/day) + active acupuncture (30 min /every day).
  Interventions: Drug: Diclectin; Device: Active acupuncture
- Diclectin plus sham acupuncture (Other): Diclectin (combination of doxylamine succinate (10 mg) and pyridoxine hydrochloride (10 mg), 2-4 tablets/day) + sham acupuncture (30 min /every day).
  Interventions: Drug: Diclectin; Device: Sham acupuncture
- Placebo plus active acupuncture (Other): Diclectin placebo (2-4 tablets/day) + active acupuncture (30 min / every day)
  Interventions: Drug: Diclectin placebo; Device: Active acupuncture
- Placebo plus sham acupuncture (Other): Diclectin placebo (2-4 tablets/day) + sham acupuncture (30 min /every day)
  Interventions: Drug: Diclectin placebo; Device: Sham acupuncture

INTERVENTIONS:
Drug: Diclectin — Diclectin (combination of 10 mg doxylamine and 10 mg pyridoxine hydrochloride in a delayed release tablet) During the first two days, patients will start with an initial oral dose of 2 tablets at bedtime. If the symptoms assessed on the second day are not relieved, 3 tablets will be administered on the third day (1 tablet in the morning and 2 tablets at bedtime). On the third day if the symptoms are still not relieved, another tablet will be added in the afternoon on the fourth day (1 tablet in the morning, 1 tablet in the afternoon and 2 tablets at bedtime). Therefore, the maximum assigned dosage of Diclectin or placebo tablets do not exceed 4 tablets per day. The treatment duration will lasts for 14 days.
  Arms: Diclectin plus active acupuncture; Diclectin plus sham acupuncture
Drug: Diclectin placebo — Diclectin placebo will be packed and tested by a commercial pharmacy supply company specifically for this study. It have the same appearance, size, batch, odor, and taste compared with Diclectin. During the first two days, patients will start with an initial oral dose of 2 tablets at bedtime. If the symptoms assessed on the second day are not relieved, 3 tablets will be administered on the third day (1 tablet in the morning and 2 tablets at bedtime). On the third day if the symptoms are still not relieved, another tablet will be added in the afternoon on the fourth day (1 tablet in the morning, 1 tablet in the afternoon and 2 tablets at bedtime). Therefore, the maximum assigned dosage of placebo tablets do not exceed 4 tablets per day. The treatment duration will lasts for 14 days.
  Arms: Placebo plus active acupuncture; Placebo plus sham acupuncture
Device: Active acupuncture — Participants will receive active acupuncture every day for 2 consecutive weeks, a total of 14 sessions. The needle will be left for 30 minutes. After de qi induced by acupuncture, the paired electrodes of the electroacupuncture device will be connected to the needle handle horizontally (except for PC6).
  Arms: Diclectin plus active acupuncture; Placebo plus active acupuncture
Device: Sham acupuncture — Blunt-tipped placebo needles will be used. Participants will receive sham acupuncture every day for 2 consecutive weeks, a total of 14 sessions. The needle will be left for 30 minutes. After de qi induced by acupuncture, the paired electrodes of the electroacupuncture device will be connected to the needle handle horizontally (except for PC6). Then, the paired electrodes of the electroacupuncture device will be connected to the needle handle horizontally (except for PC6).
  Arms: Diclectin plus sham acupuncture; Placebo plus sham acupuncture

SUMMARY:
Nausea and vomiting in pregnancy (NVP) is one of the most common symptoms of pregnancy affecting 50-85% of women during the first half of pregnancy. Maternal morbidity is common and includes psychological effects, financial burden, clinical complications from nutritional deficiencies, gastrointestinal trauma, and in rare cases, neurological damage. As the main means of alternative treatment, economical and easy to obtain; the clinical efficacy of acupuncture treatment of this disease has low level of evidence and needs to be reconfirmed. Doxylamine vitamin B6 sustained release tablets (Diclectin, combination of doxylamine succinate (10mg) and pyridoxine hydrochloride (10mg) are The American College of Obstetricians and Gynecologists recommends with Level A evidence the use of vitamin B6 in combination with doxylamine as first-line pharmacotherapy for treatment of NVP. The efficacy and safety of Diclectin has been confirmed in many years of research, but there is no evidence of high-level evidence-based medicine for the Chinese population. The purpose of this multicenter, randomized, double-blind, placebo-controlled trial was to investigate the efficacy and safety of acupuncture versus Diclectin in the treatment of NVP. We hypothesis that: (1)Sham acupuncture and Diclectin (Arm B) is more effective than sham acupuncture and placebo (Arm D); (2)Active acupuncture and placebo (Arm C) is more effective than sham acupuncture and placebo (Arm D); (3) There is no interaction (either synergistic or antagonistic effects) between the two interventions of active acupuncture and Diclectin in patients with NVP.

DETAILED DESCRIPTION:
Subjects will be randomized into one of the four treatment arms: A) active acupuncture (30 min /every day) + Diclectin (combination of doxylamine succinate (10 mg) and pyridoxine hydrochloride (10 mg) , 2-4 tablets/day); B) sham acupuncture (30 min /every day) + Diclectin (2-4 tablets/day); C) active acupuncture (30 min / every day) + Diclectin placebo (2-4 tablets/day); D) sham acupuncture (30 min /every day) + Diclectin placebo (2-4 tablets/day). Participants will receive active acupuncture or sham acupuncture treatment daily, 14 times in total, and receive Diclectin or placebo treatment every day (2 tablets at bedtime for the first two days, if the symptoms are unrelieved, add one tablet in the morning, if the symptoms are still unrelieved, add another one tablet at three o 'clock in the afternoon) for 2 consecutive weeks, 28-56 tablets in total. Daily measurement PUQE score, Visual analog scale (VAS), Adverse events and concomitant medications. Weekly visits will include global assessment of well being, adverse events and concomitant medications. The visit after treatment will assess NVP quality of life (NVPQoL), SAS, SDS and so on. Participants will be followed up 30 days after treatment. Primary outcomes is difference of the mean change in PUQE score from baseline to the last visit. Secondary outcomes were some core outcome set for hyperemesis gravidarum, including weight difference, quality of life (change in Global assessment of well-being, NVPQOL, VAS, SDS and SAS), pregnancy complication, treatment compliance, neonatal outcomes; area under the curve of PUQE score, effect of intervention on PUQE score reduction over treatment period and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Women with 20-45 years of age;
2. PUQE score ≥6;
3. 7-14 weeks of gestation with viable fetus inside the uterine cavity confirmed by ultrasound dating;
4. Less than 20% weight loss.

Exclusion Criteria:

1. Having major medical problems such as malignant tumor, acute or subacute severe hepatitis, severe aplastic anemia, idiopathic thrombocytopenic purpura, acute appendicitis, acute pancreatitis, TORCH syndrome, etc
2. Having chronic medical conditions such as poorly controlled diabetes, coronary heart disease, uncontrolled hypertension, etc
3. Coexistence of other diseases that cause vomiting such as infectious disease, gestational trophoblastic disease, etc
4. Having asthma, increased intraocular pressure, narrow-angle glaucoma, narrow peptic ulcer, pyloric obstruction, bladder neck obstruction, etc
5. Taking antiemetics such as vitamin B6, ondansetron, metoclopramide, prednisone, anti-vomiting Chinese medicine, etc., within the past week
6. Receiving conservative treatment such as dietary and lifestyle modification
7. Abnormal physical examination and laboratory tests (minor abnormalities in laboratory tests due to pregnancy vomiting, such as liver function and ions, are acceptable for inclusion)
8. Having mental handicaps or psychological disorders
9. Allergic to doxylamine, other ethanolamine-derived antihistamines, pyridoxine hydrochloride, or any inactive ingredient in diclectin
10. Using monoamine oxidase inhibitors
11. Driving or operating heavy machinery
12. Using alcohol or other central nervous system inhibitors

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 352 (Actual)
Dates: Start 2020-06-21 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Score change of pregnancy unique quantification of emesis (PUQE) scale from baseline to day 15 | Baseline to day 15; Scores ranged 3 to 15, with higher scores indicating more
  Score change of pregnancy unique quantification of emesis (PUQE) scale from baseline to day 15

SECONDARY OUTCOMES:
Score change of maternal weight from baseline to the last visit | Baseline to day 15; no range of variation
  Score change of maternal weight from baseline to the last visit
Change of electrolyte index (sodium) | Baseline to day 15
  Value changes from baseline to last Visit. Unit: mmol/L
Change of electrolyte index (potassium) | Baseline to day 15
  Value changes from baseline to last Visit. Unit: mmol/L
Change of electrolyte index (calcium) | Baseline to day 15
  Value changes from baseline to last Visit. Unit: mmol/L
Change of electrolyte index (chlorine) | Baseline to day 15
  Value changes from baseline to last Visit. Unit: mmol/L
Change of electrolyte index (phosphorus) | Baseline to day 15
  Value changes from baseline to last Visit. Unit: mmol/L
Change of electrolyte index (magnesium) | Baseline to day 15
  Value changes from baseline to last Visit. Unit: mmol/L
Change of electrolyte index (iron) | Baseline to day 15
  Value changes from baseline to last Visit. Unit: μmol/L
Change of electrolyte index (zinc) | Baseline to day 15
  Value changes from baseline to last Visit. Unit: μmol/L
Change of AST | Baseline to day 15
  Value changes from baseline to last Visit. Unit: U/L
Change of ALT | Baseline to day 15
  Value changes from baseline to last Visit. Unit: U/L
Change of ALP | Baseline to day 15
  Value changes from baseline to last Visit. Unit: U/L
Change of creatinine | Baseline to day 15
  Value changes from baseline to last Visit. Unit: μmol/L
Change of urea | Baseline to day 15
  Value changes from baseline to last Visit. Unit: mmol/L
Change of TSH | Baseline to day 15
  Value changes from baseline to last Visit. Unit: mIU/L
Change of free triiodothyronine | Baseline to day 15
  Value changes from baseline to last Visit. Unit: pmol/L
Change of free thyroxine | Baseline to day 15
  Value changes from baseline to last Visit. Unit: pmol/L
Change of vitamin b1 | Baseline to day 15
  Value changes from baseline to last Visit. Unit: ng/ml
Change of vitamin b6 | Baseline to day 15
  Value changes from baseline to last Visit. Unit: ng/ml
Change of vitamin b12 | Baseline to day 15
  Value changes from baseline to last Visit. Unit: ng/ml
Change of cortisol | Baseline to day 15
  Value changes from baseline to last Visit. Unit: ug/dL
Change of ghrelin | Baseline to day 15
  Value changes from baseline to last Visit. Unit: ng/ml
Change of leptin | Baseline to day 15
  Value changes from baseline to last Visit. Unit: ng/ml
Change of 5-hydroxytryptamine | Baseline to day 15
  Value changes from baseline to last Visit. Unit: ng/ml
Change of substance P | Baseline to day 15
  Value changes from baseline to last Visit. Unit: pg/ml
Change of arginine vasopressin plasma | Baseline to day 15
  Value changes from baseline to last Visit. Unit: pg/ml
Change of GDF 15 | Baseline to day 15
  Value changes from baseline to last Visit. Unit: pg/ml
Change of IGFBP 7 | Baseline to day 15
  Value changes from baseline to last Visit. Unit: ng/ml
Intravenous fluid treatment during treatment | Baseline to day 15
  Intravenous fluid treatment during treatment
Concomitant treatment | Baseline to day 15
  Concomitant treatment
Hospital admission during treatment | Baseline to day 15
  Hospital admission during treatment
Termination of pregnancy | Data collected from baseline to the end of follow-up period (four weeks after the end of treatment).
  Termination of pregnancy. If the patient is suffering further aggravation of hyperemesis gravidarum, the termination of a wanted pregnancy will be done due to life in danger. Or congenital anomalies are found by ultrasound, the termination of a wanted pregnancy will be done.
Maternal outcomes | Data collected from baseline to 42 days after postpartum.
  Including pregnancy complications, termination of pregnancy and birth outcomes. Pregnancy complications including miscarriage (in the first trimester and in the second trimester), hypertensive disorders, and gestational diabetes; birth outcomes including live birth, vaginal delivery, cesarean section, gestational age, preterm, birth weight and small for gestational age.
Patient satisfaction with treatment | Baseline to day 15
  Such as loss of confidence or intolerance to daily acupuncture and so on
Treatment compliance | Baseline to day 15
  Such as the percentage of drug or needle used; or drug tablets or acupuncture sessions.
Offspring outcomes | Data collected from baseline to to 42 days after postpartum.
  Including fetal and neonatal congenital anomalies, fetal and neonatal mortality, neonatal hypoglycemia and NICU admission.
Area under the curve (AUC) of PUQE score over treatment | Baseline to day 15
  Scores ranged 3 to 15, with higher scores indicating more severe NVP
PUQE score reduction based on different TCM patterns | Scores ranged 3 to 15, with higher reduction indicating the better
  PUQE score reduction based on different TCM patterns
Adverse events and serious adverse events | Baseline to the end of follow-up (four weeks after the end of treatment)
  The percentage of adverse events and serious adverse events
Quality of life: NVPQoL | Baseline to day 15
  Range 30-210, high being poor QoL
Quality of life: VAS | Baseline to day 15
  Ranged 0-10, high being more severe symptoms
Quality of life: SDS | Baseline to day 15
  Range 25-10, high being more severe
Quality of life: SAS | Baseline to day 15
  Range 25-100, high being more severe
Quality of life: global assessment of well-being | Baseline to day 15
  Range 0-10, low being more severe
PUQE score reduction at different levels of NVP | Scores ranged 3 to 15, with higher reduction indicating the better
  PUQE score reduction at different levels of NVP

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoke Wu, Ph.D, Study Chair — First Affiliated Hospital of Heilongjiang University of Chinese Medicine
Locations (13):
- China (13):
  - First Affiliated Hospital of Heilongjiang Chinese Medicine University, Harbin, Heilongjiang
  - Heilongjiang provincial hospital, Harbin, Heilongjiang
  - Hegang Maternal and Child Health Hospital, Hegang, Heilongjiang
  - Affiliated Hospital of Jiamusi Medical University, Jiamusi, Heilongjiang
  - Jiamusi Maternal and Child Health Hospital, Jiamusi, Heilongjiang
  - Jixi Maternal and Child Health Hospital, Jixi, Heilongjiang
  - Mudanjaing Maternal and Child Health Hospital, Mudanjiang, Heilongjiang
  - Shuangyashan Maternal and Child Health Hospital, Shuangyashan, Heilongjiang
  - Suihua Maternal and Child Health Hospital, Suihua, Heilongjing
  - Luoyang Hospital of TCM, Luoyang, Henan
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Ningxia Hui Autonomous Region Hospital of TCM, Yinchuan, Ningxia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu XK, Gao JS, Ma HL, Wang Y, Zhang B, Liu ZL, Li J, Cong J, Qin HC, Yang XM, Wu Q, Chen XY, Lu ZL, Feng YH, Qi X, Wang YX, Yu L, Cui YM, An CM, Zhou LL, Hu YH, Li L, Cao YJ, Yan Y, Liu L, Liu YX, Liu ZS, Painter RC, Ng EHY, Liu JP, Mol BWJ, Wang CC. Acupuncture and Doxylamine-Pyridoxine for Nausea and Vomiting in Pregnancy : A Randomized, Controlled, 2 x 2 Factorial Trial. Ann Intern Med. 2023 Jul;176(7):922-933. doi: 10.7326/M22-2974. Epub 2023 Jun 20. PMID 37335994